CLINICAL TRIAL: NCT03723551
Title: Randomized Open-label Active-controlled Study to Assess the Safety, Tolerability, and Efficacy of Afabicin IV/Oral in the Treatment of Patients With Bone or Joint Infection Due to Staphylococcus
Brief Title: Study to Assess Safety, Tolerability and Efficacy of Afabicin in The Treatment of Participants With Bone or Joint Infection Due to Staphylococcus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial was concluded for strategic reasons.
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1450-BJI-205
Record Dates: First submitted 2018-10-26; First posted 2018-10-29 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Bone or Joint Infection
MeSH Terms: interventions — afabicin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afabicin (Experimental): In Part A, afabicin will be given intravenous (IV) at a dose 160 milligrams (mg) twice daily (BID) for a minimum of 1 day (at least 1 dose) and up to a maximum of 14 days (2 weeks), followed by a switch to oral Afabicin at a dose of 240 mg BID for the remaining treatment duration.
  In Part B, participants will be administered with open label afabicin IV at a dose of 55 mg BID for a minimum of 1 day (at least 1 dose) and up to a maximum of 14 days (2 weeks) followed by a switch to oral afabicin at a dose of 80 mg BID for the remaining treatment duration. In certain study conditions a higher dosing regimen of afabicin might be used: afabicin intravenous (IV) at a dose of 80 mg BID for a minimum of 1 day (at least 1 dose) and up to a maximum of 14 days (2 weeks) followed by a switch to oral afabicin at a dose of 120 mg BID for the remaining treatment duration.
  Interventions: Drug: Afabicin
- Standard of Care (SOC) (Parts A and B) (Active Comparator): Participants will be administered with SOC in accordance with local practice and applicable treatment guidelines without exceeding the maximum dosing schedule.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Afabicin — Administered intravenously and orally.
  Arms: Afabicin
Drug: Standard of Care — Administered with SOC in accordance with local practice and applicable treatment guidelines.
  Arms: Standard of Care (SOC) (Parts A and B)

SUMMARY:
This is a randomized, active-controlled, open-label study to assess the safety, tolerability and efficacy of Afabicin in the treatment of participants with bone or joint infection due to Staphylococcus aureus [both methicillin-susceptible S. aureus (MSSA) and methicillin-resistant S. aureus (MRSA)] and/or coagulase-negative staphylococci (CoNS) and to compare it to standard of care (SOC).

ELIGIBILITY:
Key Inclusion Criteria:

* Able to provide written informed consent and to comply with study procedures.
* Diagnosis of bone or joint infection which fulfils the following conditions: a) Infection is due to S. aureus (MSSA or MRSA) and/or CoNS only; and, b) Participants had received no more than 7 days of empiric antibiotics prior to initiating treatment with study drug unless the pathogen isolated was resistant to the administered empiric antibiotics; and, c) Biofilm is not considered to be yet established and/or has been mechanically eradicated; and, d) Infection is not associated with an ischiatic or a sacral osteomyelitis; and e) Infection can involve periosteal or soft tissue.

Key Exclusion Criteria:

* Presence of co-infection with non-staphylococcal bacteria at the affected joint or bone site, or in the blood.
* Participants at an increased risk of developing liver injury.
* Participants who have medical conditions that increase the risk of QT prolongation.
* Medical history within the previous 3 months of: myocardial infarction, unstable angina pectoris, coronary artery or cerebral revascularization procedure or stroke, ventricular tachycardia, multifocal ventricular ectopics requiring treatment, or any other clinically relevant symptomatic ventricular arrhythmias.
* Documented history of alcohol or drug abuse within the previous 12 months.
* For patients with DFO:

  1. Severe peripheral arterial disease (PAD) requiring revascularization; however, patients with peripheral artery disease are eligible for inclusion, provided they have undergone successful revascularization or it has been deemed unnecessary by a vascular surgeon
  2. Necrotizing fasciitis or gangrene requiring complete lower extremity amputation (of all infected bone and soft tissue).
  3. Patients with Charcot foot (suspected neuro-osteoarthropathy according to Investigator's judgment).
  4. Need for digital amputation.
* Life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) Based on Nature, Incidence, Severity, Seriousness, and Outcome | Baseline up to 12-weeks post- end of treatment (EOT)
Change from Baseline in Number of Participants With Incidence of Laboratory Abnormalities | Baseline up to Week 12 post- EOT

SECONDARY OUTCOMES:
Proportion of Participants With Clinical Response | Days 8, 28, 42, EOT, 4-weeks and 12-weeks post- EOT, as applicable up to Day 168

CONTACTS AND LOCATIONS:
Locations (19):
- Georgia (7):
  - Georgian Clinics JSC, Akhalts'ikhe
  - West Georgia Medical Center LLC, Kutaisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center LLC, Tbilisi
  - LEPL The First University Clinic of Tbilisi State Medical University, Tbilisi
  - Tbilisi State Medical University And Ingorokva High Medical Technology University Clinic LLC, Tbilisi
  - Academician Vakhtang Bochorishvili Clinic LTD, Tbilisi
  - Caucasus Medical Center LLC, Tbilisi
- South Africa (3):
  - Worthwhile Clinical Trials, Lakeview Hospital, Benoni
  - Clinical Research Unit, University of Pretoria, Pretoria
  - Global Clinical Trials (Pty) Ltd, Pretoria
- Ukraine (9):
  - Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - Regional Clinical Hospital under Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Kharkiv Regional Clinical Traumatology Hospital, Kharkiv
  - Institute of Traumatology and Orthopedics, Kyiv
  - Kyiv Regional Clinical Hospital, Kyiv
  - Kyiv City Clinical Hospital #8 under the Executive Body of Kyiv City Council (Kyiv City State Administration), Kyiv
  - Vinnytsya Regional Clinical Hospital, Vinnytsia
  - Lviv Regional Hospital of Veterans of Wars and Repressed after Yurii Lypa, Vynnyky
  - City Hospital #9 under Zaporizhia City Council, Zaporizhia